CLINICAL TRIAL: NCT05024071
Title: Effect of Core Strength Training on C-level Difficulty Movements of Wushu Routine Athletes
Brief Title: Effect of Core Strength Training on Wushu C-level Difficulty Movements ,12 Weeks of Core Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Li Long, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: Li Long
Record Dates: First submitted 2021-08-09; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Experimental Myasthenia
Keywords: Core strength training; C-level difficulty; Wushu routine
MeSH Terms: conditions — Myasthenia Gravis, Autoimmune, Experimental

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swiss Ball (Experimental): Swiss ball practice can create an unstable environment, promote the recovery of muscle function and develop joint stability. It can train the muscle groups in chest, abdomen, back, buttocks and legs, which play an important role in maintaining body balance and improving athletes' body.
  Interventions: Device: Wushu athletes in the experimental group used a Swiss ball for 12 weeks of core strength training; Device: Wushu athletes in the experimental group used a balance board for 12 weeks of core strength training
- Balance Plate (Experimental): The balance board can exercise athletes' waist explosive force and body balance ability in an unstable state.
  Interventions: Device: Wushu athletes in the experimental group used a Swiss ball for 12 weeks of core strength training; Device: Wushu athletes in the experimental group used a balance board for 12 weeks of core strength training

INTERVENTIONS:
Device: Wushu athletes in the experimental group used a Swiss ball for 12 weeks of core strength training — The experimental group was given 12 weeks of core strength training, divided into 6 types
  1. Static action under steady state.
  2. No load movement in steady state.
  3. Static action under unstable state.
  4. Movement to overcome its own resistance in an unstable state.
  5. Free strength exercise in unstable state.
  6. Core explosive power exercise under unstable conditions.
Device: Wushu athletes in the experimental group used a balance board for 12 weeks of core strength training — The experimental group was given 12 weeks of core strength training, divided into 6 types
  1. Static action under steady state.
  2. No load movement in steady state.
  3. Static action under unstable state.
  4. Movement to overcome its own resistance in an unstable state.
  5. Free strength exercise in unstable state.
  6. Core explosive power exercise under unstable conditions.

SUMMARY:
This paper designs the core strength training scheme based on the query and reference of relevant literature and the characteristics of C-level difficult movements of Wushu. The training plan of the experimental group includes three stages (weeks 1-3; weeks 4-9; and week 10-12). Each stage consists of different difficulty levels. The training program is divided into 6 difficulty levels.

DETAILED DESCRIPTION:
Effect of core strength training on C-level difficulty movements of Wushu routine athletes Dear Professor Hello! Investigator, a doctoral student in physical education at UPM. This is an experimental research process on the impact of core strength training on the C- level difficulty of Competitive Wushu routines. The subjects were 18-22 year old Wushu athletes. The data obtained from this survey are only for academic research. Therefore,investigator sincerely invite experts to score each stage of investigator experiment, help investigator do this experiment better. Thank you very much.

This paper designs the core strength training scheme based on the query and reference of relevant literature and the characteristics of C-level difficult movements of Wushu. The training plan of the experimental group includes three stages (weeks 1-3; weeks 4-9; and week 10-12). Each stage consists of different difficulty levels. The specific training contents are as follows:

Core Strength Training Plan. (Weeks 1-3; weeks 4-9; and weeks 10-12)

1. Basic stage of core strength training Training time: 30 minutes three times a week for 1-3 weeks Training content: static action in stable state, no-load movement in stable state and static action in unstable state Number and times of training groups Contents of core strength training in week 1-3 basic stage Training Phase Training Content Time And Frequency Preparation part (5 minutes) Jogging 3 minutes 3×50 m Neck movement (front, rear, left and right) 30 S 4×8 Shoulder movement 30 S 4×8 Waist movement 30 S 4×8 Lunge leg press 30 S 4×8 Static action under steady state (12 minutes) Flat brace 60 S × 2 groups Single side support of flat support (left) 60 S × 2 groups Single side support of flat support (right) 60 S × 2 groups Reverse plate support 60 S × 2 groups Side bridge elbow support (left) 60 S × 2 groups Side bridge elbow support (right) 60 S × 2 groups No load movement in steady state (9 minutes) Suspension leg lift 60 S × 3 groups Drape knees and tuck in (left) 60 S × 2 groups Drape, bend knees and tuck in (right) 60 S × 2 groups Hanging upside down 60 S × 2 groups Static action under unstable state (4 minutes) Lateral hip abduction (left) 60 S × 2 groups Lateral hip abduction (right) 60 S × 2 groups
2. Core strength training consolidation stage Training time: 30 minutes three times a week for 4-9 weeks Training content: Static action in unstable state, movement to overcome self-resistance in unstable state, free force exercise in unstable state.

   Number and times of training groups (Table 3) Table 3 contents of core strength training in week 4-9 basic stage Training Phase Training Content Time And Frequency Preparation part (6 minutes) Jogging 4 minutes 4×50 m Neck movement (front, rear, left and right) 30 S 4×8 Shoulder movement 30 S 4×8 Waist movement 30 S 4×8 Lunge leg press 30 S 4×8 Static action under unstable state (6 minutes) Lateral hip abduction (left) 60 S ×3 groups Lateral hip abduction (right) 60 S × 3 groups Movement to overcome its own resistance in an unstable state (9 minutes) Push down leg arm flat hip (left) 60 S × 3 groups Push down leg arm flat hip (right) 60 S ×3 groups Upside down abdominal retraction (bilateral) 60 S ×3 groups Free strength exercise in unstable state (9 minutes) Prone mass body 60 S × 3 groups Prone push-pull 60 S × 3 groups Swiss Ball push up 60 S × 3 groups
3. Core strength training improvement stage Training time: 30 minutes three times a week for 10-12 weeks Training contents: free strength exercise under unstable conditions, core explosive force exercise under unstable conditions, and core special strength exercise under unstable conditions.

Number and times of training groups (Table 4) Table 4 contents of core strength training in week 4-9 basic stage Training Phase Training Content Time And Frequency Preparation part (4 minutes) Jogging 2 minutes 2×50 m Neck movement (front, rear, left and right) 30 S 4×8 Shoulder movement 30 S 4×8 Waist movement 30 S 4×8 Lunge leg press 30 S 4×8 Free strength exercise in unstable state (10 minutes) Flat brace (two points) 60 S × 2 groups Prone mass body 60 S ×2 groups Prone push-pull 60 S ×2 groups Swiss Ball push up 60 S × 4 groups No load movement in steady state (8 minutes) Suspension leg lift 60 S × 2 groups Drape knees and tuck in (left) 60 S × 2 groups Drape, bend knees and tuck in (right) 60 S × 2 groups Hanging upside down 60 S × 2 groups Core explosive force exercise under non-stability (8 minutes) Lie on your back and bend your knees at both ends 60 S × 2 groups Plate support knee lift 60 S × 2 groups Rotation of stretch belt (both sides) 60 S × 2 groups Lie on your back and throw the ball 60 S × 2 groups

ELIGIBILITY:
Inclusion Criteria:

1. Wushu athlete
2. Lives in Ningxia Wushu Professional Team
3. Ages 18-22
4. The difficulty movement training has not been exposed to the core strength training

Exclusion Criteria:

1. They don't live in Ningxia
2. There are physical injuries
3. Younger than 18 years old and older than 22 years old
4. Have core strength training experience

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Basic stage of core strength training (s) | 4 weeks
  1. Static action under steady state Flat brace(s) Single side support of flat support (left) (s) Single side support of flat support (right) (s) Reverse plate support (s) Side bridge elbow support (left) (s) Side bridge elbow support (right) (s)
  2. No load movement in steady state Suspension leg lift (s) Drape knees and tuck in (left) (s) Drape, bend knees and tuck in (right) (s) Hanging upside down (s)
  3. Static action under unstable state Lateral hip abduction (left) (s) Lateral hip abduction (right) (s)
Core strength training consolidation stage (s) | 10 weeks
  1. Static action under unstable state Lateral hip abduction (left) (s) Lateral hip abduction (right) (s)
  2. Movement to overcome its own resistance in an unstable state Push down leg arm flat hip (left) (s) Push down leg arm flat hip (right) (s) Upside down abdominal retraction (bilateral) (s)
  3. Free strength exercise in unstable state Prone mass body (s) Prone push-pull (s) Swiss Ball push up (s)
Core strength training improvement stage (s) | 13 weeks
  1. Free strength exercise in unstable state Flat brace (two points) (s) Prone mass body (s) Prone push-pull (s) Swiss Ball push up (s)
  2. No load movement in steady state Suspension leg lift (s) Drape knees and tuck in (left) (s) Drape, bend knees and tuck in (right) (s) Hanging upside down (s)
  3. Core explosive force exercise under non-stability Lie on your back and bend your knees at both ends (s) Plate support knee lift (s) Rotation of stretch belt (both sides) (s) Lie on your back and throw the ball (s)

CONTACTS AND LOCATIONS:
Overall Officials: Long Li, Principal Investigator — University Putra Malaysia
Locations (1):
- Ningxia sports vocational and Technical College, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No
Because this is my doctoral thesis and it has certain confidentiality, I won't share it until I finish my doctoral thesis.

REFERENCES:
- [Result] Myer GD, Ford KR, Palumbo JP, Hewett TE. Neuromuscular training improves performance and lower-extremity biomechanics in female athletes. J Strength Cond Res. 2005 Feb;19(1):51-60. doi: 10.1519/13643.1. PMID 15705045
- See also: This article is from Google literature. — https://paulogentil.com/

DOCUMENTS (1):
  • Study Protocol (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05024071/Prot_000.pdf